CLINICAL TRIAL: NCT03241589
Title: Teledermatology Mobile Apps: Implementation and Impact on Veterans' Access to Dermatology
Brief Title: Teledermatology Mobile App: Patient Facing
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SDR 16-192
Record Dates: First submitted 2017-07-26; First posted 2017-08-07 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Introduction of Teledermatology Mobile Apps
Keywords: Teledermatology; Telehealth; Dermatology; Telemedicine; Mobile Application

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Rural Veterans: Originally the aim was to include VA sites who received the direct to patient facing app from OCC. Due to a lack of enrollment, the first arm or group has been redefined as Veterans living in rural areas receiving a request to use the patient facing app.
  Interventions: Other: Direct to patient facing mobile apps introduction
- Nonrural Veterans: Originally the comparison group consisted of VA sites to eventually receive the direct to patient facing apps. Since our enrollment at the facility level was low, this arm now consists of Veterans receiving a request to use the patient facing app, living in nonrural areas.
  Interventions: Other: Direct to patient facing mobile apps introduction

INTERVENTIONS:
Other: Direct to patient facing mobile apps introduction — VA employees and Veterans begin use of OCC's direct to patient facing mobile app.

SUMMARY:
This study was designed to measure the impact of two teledermatology apps to provide direct to patient teledermatology follow up care, Patient Viewer and My VA Images, with a trial on access to dermatology care. The overall hypothesis was that sites implementing Department of Veterans Affairs' (VA) teledermatology mobile apps would significantly augment the use of teledermatology and improve Veterans' access to skin care relative to control sites. Specifically, the investigators hypothesized that these apps would improve established patients' ability to follow-up with dermatology care remotely, reducing patient travel to dermatology clinics while opening up dermatology clinic space for other patients. Due to a lack of participation by sites during the study which was conducted during the novel coronavirus (COVID-19) pandemic, the groups examined are Veterans who live in rural areas compared to those in urban areas.

Previously the study included a parallel trial to evaluate another teledermatology mobile app, VA Telederm. This trial was no longer feasible within this study's funding timeline due to limitations imposed on the mobile app by Office of Information & Technology that were not under the control of the PI or the operational partner, Office of Connected Care (OCC).

DETAILED DESCRIPTION:
Access to healthcare is a key priority for the Department of Veterans Affairs (VA). The current practice of teledermatology in VA is effective but has not been uniformly implemented. Once patients establish care in a dermatology clinic, they often need follow-up visits to evaluate responses to treatment and to adjust management, neither of which necessarily requires a face-to-face visit. To improve clinic access to in-person dermatology clinics, VA Office of Connected Care developed a patient-facing mobile app, My VA Images, to be used in conjunction with the clinician-facing Patient Viewer app, to allow established dermatology clinic patients to follow-up remotely by submitting digital skin images and interval history. The mobile apps were planned for wide-spread implementation in the VA. The investigators conducted a trial of database review to understand how these two apps affected features of dermatology care, specifically related to access to care.

The apps were made available over a 1 year and 4 month period in a cluster randomized, stepped-wedge design to Veterans Health Administration (VHA) facilities. The direct-to-patient facing apps were distributed to 31 facilities with dermatology clinics that had recent relatively high teledermatology activity and thus already had relatively mature teledermatology programs ready for advanced operations.

By using a stop code unique to this process, the investigators planned to use the VA Corporate Data Warehouse (CDW) to measure effectiveness of the apps on all outcomes reflecting dermatology access. Due to an unexpectedly small sample size resulting from poor adoption of the intervention, in part during the COVID-19 pandemic, analysis using the cluster-randomized stepped wedge design evaluation was not warranted. Instead, we focused on understanding factors associated with successful completion of consults with the mobile apps, examining differences between rural and urban Veteran users. The results are of significance to VA as it develops and implements other mobile telehealth programs, and more generally to other healthcare organizations planning for large-scale telehealth interventions.

The planned study originally also included a parallel trial to evaluate another teledermatology mobile app, VA Telederm, designed to facilitate adoption of consultative teledermatology and enhance overall access to dermatology opinion in VA. Unforeseen changes in the app hosting environment imposed by VA Office of Information and Technology early in the study and not under the control of the PI or the operational partner, Office of Connected Care (OCC), rendered the app non-functional, and the trial was no longer feasible within this study's funding timeline were not under the control of the PI or the operational partner, Office of Connected Care (OCC). Organizational readiness for change for the VA Telederm app was measured.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion for the trial with direct to patient facing apps was that a site had greater than or equal to 9% of all Fiscal Year (FY) 2018 dermatology encounters under secondary stop codes 695/696.
* This indicated considerable pre-existing experience with consultative teledermatology and the likely presence of dermatology reader and support personnel needed to implement direct to patient facing apps.
* The investigators identified 31 sites eligible for direct to patient facing apps.
* We followed above criteria but due to low enrollment, an additional criteria was added that patients were included if they received a request to use the patient-facing mobile app.

Exclusion Criteria:

* VA medical centers with no 695/696 stop code activity in FY2018 or with zero full-time equivalent dermatologists were excluded since these sites likely lacked the expertise, support, and infrastructure to feasibly adopt teledermatology during the study period.
* The investigators also excluded sites outside the continental U.S., and sites without a dermatology clinic.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients at sites in study who received consultative teledermatology requests via My VA Images.
Sampling Method: Non-Probability Sample
Enrollment: 466 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis H. Oh, MD PhD, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (3):
- United States (3):
  - San Francisco VA Medical Center, San Francisco, CA, San Francisco, California
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peracca SB, Jackson GL, Jackson MA, Oh DH. Implementation of Teledermatology: Theory and Practice. Current Dermatology Reports. 2019 Jun 1; 8(2):35-45.
- [Result] Done N, Oh DH, Weinstock MA, Whited JD, Jackson GL, King HA, Peracca SB, Elwy AR, Prentice JC. VA Telederm study: protocol for a stepped-wedge cluster randomised trial to compare access to care for a mobile app versus a workstation-based store-and-forward teledermatology process. BMJ Open. 2018 Dec 14;8(12):e022218. doi: 10.1136/bmjopen-2018-022218. PMID 30552249
- [Result] Fonseca A, Peracca SB, Lachica O, Morris I, King H, Jackson G, Whited J, Oh DH, Weinstock MA. 379 Implementing a teledermatology patient-facing mobile application in the VA. [Abstract]. The Journal of Investigative Dermatology. 2020 Jul 1; 140(7):S48.
- [Result] Peracca S, Fonseca A, Grenga A, Jackson G, King H, Chapman J, Whited J, Weinstock M, Oh DH. 411 Implementation of a consultative teledermatology mobile application in Veterans Affairs. [Abstract]. The Journal of Investigative Dermatology. 2020 Jul 1; 140(7):S53.
- [Result] Peracca SB, Fonseca A, Hines A, King HA, Grenga AM, Jackson GL, Whited JD, Chapman JG, Lamkin R, Mohr DC, Gifford A, Weinstock MA, Oh DH. Implementation of Mobile Teledermatology: Challenges and Opportunities. Telemed J E Health. 2021 Dec;27(12):1416-1422. doi: 10.1089/tmj.2020.0500. Epub 2021 Mar 1. PMID 33691074
- [Result] Lewinski AA, Crowley MJ, Miller C, Bosworth HB, Jackson GL, Steinhauser K, White-Clark C, McCant F, Zullig LL. Applied Rapid Qualitative Analysis to Develop a Contextually Appropriate Intervention and Increase the Likelihood of Uptake. Med Care. 2021 Jun 1;59(Suppl 3):S242-S251. doi: 10.1097/MLR.0000000000001553. PMID 33976073
- [Derived] Peracca SB, Lachica O, Lamkin RP, Jackson GL, Mohr DC, King HA, Whited JD, Fonseca AS, Morris IJ, Gifford AL, Weinstock MA, Oh DH. Implementation of Direct-to-Patient Mobile Teledermatology in VA. J Gen Intern Med. 2024 Feb;39(Suppl 1):97-105. doi: 10.1007/s11606-023-08480-1. Epub 2024 Jan 22. PMID 38252250
- [Derived] Peracca SB, Fonseca AS, Lachica O, Jackson GL, Morris IJ, King HA, Misitzis A, Whited JD, Mohr DC, Lamkin RP, Gifford AL, Weinstock MA, Oh DH. Organizational Readiness for Patient-Facing Mobile Teledermatology to Care for Established Veteran Patients in the United States. Telemed J E Health. 2023 Jan;29(1):72-80. doi: 10.1089/tmj.2022.0009. Epub 2022 May 24. PMID 35612465

RESULTS

PARTICIPANT FLOW:
Groups:
- Rural Veterans: Originally the aim was to include VA sites who received the direct to patient facing app from Office of Connected Care (OCC). Due to a lack of enrollment, the first arm or group has been redefined as Veterans living in rural areas.
  Direct to patient facing mobile apps introduction: VA employees and Veterans begin use of OCC's direct to patient facing mobile app. The two arms occur simultaneously.
- Nonrural Veterans: Originally VA sites to eventually receive the direct to patient facing apps but at present had not were in the second arm or control group. Since our enrollment at the facility level was low, this arm now consists of Veterans living in nonrural areas.
  Direct to patient facing mobile apps introduction: VA employees and Veterans begin use of OCC's direct to patient facing mobile app. The two arms occur simultaneously.
Period: Overall Study
Arm/Group | Rural Veterans | Nonrural Veterans
Started | 109 | 357
Completed | 109 | 357
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population is all Veteran patients who were given the opportunity to use the My VA Images app.
Groups:
- Rural Veterans: Originally the aim was to include VA sites who received the direct to patient facing app from OCC. Due to a lack of enrollment, the first arm or group has been redefined as Veterans living in rural areas.
  Direct to patient facing mobile apps introduction: VA employees and Veterans begin use of OCC's direct to patient facing mobile app. The two arms occur simultaneously.
- Total: Total of all reporting groups
Arm/Group | Rural Veterans | Nonrural Veterans | Total
Number analyzed (Participants) | 109 | 357 | 466
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 189 | 222
  >=65 years | 76 | 168 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.31 (12.10) | 61.54 (14.83) | 62.89 (14.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 61 | 71
  Male | 99 | 296 | 395
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 10 | 12
  Not Hispanic or Latino | 103 | 332 | 435
  Unknown or Not Reported | 4 | 15 | 19
Region of Enrollment [Number; unit: participants]
  United States | 109 | 357 | 466

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants That Successfully Completed Remote Follow up
Description: Whether patient had a successful completion of a remote follow-up visit during the study period, which included 1 year and 4 months. The time frame of the follow up varied as clinically appropriate.
Time Frame: 1 year 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Rural Veterans: Originally the aim was to include VA sites who received the direct to patient facing app from OCC. Due to a lack of enrollment, the first arm or group has been redefined as Veterans with living in rural areas.
  Direct to patient facing mobile apps introduction: VA employees and Veterans begin use of OCC's direct to patient facing mobile app.
- Nonrural Veterans: Originally VA sites to eventually receive the direct to patient facing apps but at present had not were in the second arm or control group. Since our enrollment at the facility level was low, this arm now consists of Veterans living in nonrural areas.
  Direct to patient facing mobile apps introduction: VA employees and Veterans begin use of OCC's direct to patient facing mobile app.
Arm/Group | Rural Veterans | Nonrural Veterans
Number analyzed (Participants) | 109 | 357
Participants | 51 | 182
Statistical Analysis 1: Comparison: Rural Veterans vs Nonrural Veterans; We followed power calculations described in uploaded protocol document, using an incomplete design matrix with a 3-month transition period, a level of precision α=0.05 and a minimum power level of 0.80. We also assumed a total number of clusters I=36 as per the study design and the number of baseline measurements B=2. Due to insufficient sample size, we modified groups studied; Test type: Superiority; p = 0.7428, Regression, Logistic; Odds Ratio (OR) = 0.931, 95% CI 2-sided [0.606 to 1.429] — Referent group is Urban

2. Primary Outcome: Total Number of Participants Who Ever Completed Remote Follow-up Requests
Description: Ever completed is defined as those who at first experienced an expired request or no show but eventually completed the request, after subsequent requests were submitted for the same problem. The time frame for the follow-up of each patient was clinically appropriate determined by the dermatologist and thus varied. The collection of whether or not the follow up of patients were ever completed took place over the study period of 1 year and 4 months.
Time Frame: 1 year 4 months
Population: Users of a direct-to-patient facing mobile app at participating sites.
Measure: Count of Participants; unit: Participants
Groups:
- Rural Veterans: The first group is defined as Veterans living in rural areas receiving a request to use the patient facing app.
- Nonrural Veterans: This group consists of Veterans receiving a request to use the patient facing app, living in nonrural areas.
Arm/Group | Rural Veterans | Nonrural Veterans
Number analyzed (Participants) | 109 | 357
Participants | 18 | 30
Statistical Analysis 1: Comparison: Rural Veterans vs Nonrural Veterans; Test type: Superiority; p = 0.0031, Regression, Logistic; 2 degrees of freedom, Wald Chi-Square 11.5759; Odds Ratio (OR) = 2.258, 95% CI 2-sided [1.181 to 4.315] — Veterans with expired requests = referent

ADVERSE EVENTS:
Time Frame: 5/13/2019-9/30/2020 1 1/2 years, over the entire study period. The study did not intervene in clinical practice but reviewed the data administratively. Adverse events for specific patients were reviewed operationally by appropriate clinical staff, the study reviewed if any adverse events took place over the course of the study.
Description: All-cause mortality was not monitored and thus data are not available.
Groups:
- Rural Veterans: Rural Veterans use of OCC's direct to patient facing mobile app.
  Originally the aim was to include VA sites who received the direct to patient facing app from OCC. Due to a lack of enrollment, the first arm or group has been redefined as Veterans living in rural areas.
- Nonrural Veterans: Nonrural Veterans use of OCC's direct to patient facing mobile app.
  Originally VA sites to eventually receive the direct to patient facing apps but at present had not were in the second arm or control group. Since our enrollment at the facility level was low, this arm now consists of Veterans living in nonrural areas.
Arm/Group | Rural Veterans | Nonrural Veterans
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/357
Other Adverse Events (participants affected / at risk) | 0/109 | 0/357

LIMITATIONS AND CAVEATS:
Due to an unexpectedly small sample size resulting from poor adoption of the intervention by sites during the study, which was in part conducted during the novel coronavirus (COVID-19) pandemic, we were not able to follow the original cluster-randomized stepped wedge analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT03241589/Prot_SAP_000.pdf